CLINICAL TRIAL: NCT05312125
Title: Comparison of the Effectiveness of Different Physiotherapy and Rehabilitation Programs After Onabotulinum Toxin-A Injection and Serial Casting in Children With Cerebral Palsy
Brief Title: Physiotherapy After Botulinum Toxin Injection and Serial Casting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Gulhane Training and Research Hospital (Other Government); Ankara Eğitim ve Araştırma Hastanesi (Unknown)
Responsible Party: Principal Investigator, pelin atalan, Physiotherapist, MSc, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GaziUniPA
Record Dates: First submitted 2022-03-08; First posted 2022-04-05 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cerebral Palsy; Cerebral Palsy, Spastic
Keywords: cerebral palsy; botulinum toxin; serial casting; physiotherapy; muscle morphology
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: 2 groups of children with Cerebral palsy are going to be involved at the same time. One of the groups will be enrolled in the routine physiotherapy intervention. The other group will be enrolled to the routine physiotherapy intervention + backward downhill walking.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Children in this group will take routine physiotherapy (stretching, strengthening) program during 6 weeks. 3 days/week.
  Interventions: Procedure: routine physiotherapy
- intervention group (Active Comparator): Children in this group will take routine physiotherapy (stretching, strengthening) program + backward downhill walking (10 minutes in a day) during 6 weeks. 3 days/week.
  Interventions: Procedure: backward downhill walking; Procedure: routine physiotherapy

INTERVENTIONS:
Procedure: backward downhill walking — Children in the intervention group will take backward downhill walking program plus to routine physiotherapy.
  Arms: intervention group
Procedure: routine physiotherapy — Children in one of the groups will take routine physiotherapy programme

SUMMARY:
The effects of different physiotherapy programs on children with cerebral palsy who have been received botulinum toxin injection and serial casting application will be determined.

DETAILED DESCRIPTION:
CP children who underwent botulinum toxin injection to medial gastrocnemius muscle and serial casting application in last two months will be included in the study. The effects of traditional physiotherapy and downhill backward treadmill training plus to traditional physiotherapy on muscle morphology, activity, walking, quality of life and selectivity will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with cerebral palsy (CP) (hemiplegic-diplegic)
2. To have undergone botulinum toxin and serial casting interventions in the last 2 months
3. to be between 5-10 years old
4. Being at the level of I-II-III (ambulatory or assisted ambulatory) according to Gross Motor Function Classification System
5. To have the mental competence to understand and apply assessments and exercises

Exclusion Criteria:

1. Having undergone surgery involving the lower extremity in the last 6 months
2. Refusing to participate in the study
3. Having other accompanying neurometabolic or orthopedic disorders

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Muscle morphology | Before the intervention
  Muscle thickness, cross sectional area, fiber length, pennation angle will be recorded by ultrasonographic measurements
Muscle morphology | After six weeks intervention
  Muscle thickness, cross sectional area, fiber length, pennation angle will be recorded by ultrasonographic measurements
Vascularization | Before the the intervention
  Muscle vascularization will be recorded by Suberb Microvascular Imaging (SMI) method via ultrasonographic measurements
Vascularization | After six weeks intervention
  Muscle vascularization will be recorded by Suberb Microvascular Imaging (SMI) method via ultrasonographic measurements
Muscle strenght | Before the intervention
  Will be measured by manual muscle tester
Muscle strenght | After six weeks intervention
  Will be measured by manual muscle tester
Range of motion | Before the intervention.
  Will be measured with goniometer
Range of motion | After six weeks intervention
  Will be measured with goniometer
Edinburgh visual gait analysis | Before the intervention
  Gait will be recorded as video and this video will be scored
Edinburgh visual gait analysis | After six weeks intervention
  Gait will be recorded as video and this video will be scored
Modified Tardieu Scale | Before the intervention
  Lower extremity spasticity will be mesured with this scale. Higher scores mean more intensive spasticity
Modified Tardieu Scale | After six weeks intervention
  Lower extremity spasticity will be mesured with this scale. Higher scores mean more intensive spasticity

SECONDARY OUTCOMES:
Demographic data | Before the intervention
  Face-to-face interview with family. Will be recorded in data registration form
Demographic data | After six weeks intervention
  Face-to-face interview with family. Will be recorded in data registration form
Child Health Questionnare (Parent form) | Before the intervention
  Quality of life will be measured by this questionnare
Child Health Questionnare (Parent form) | After six weeks intervention
  Quality of life will be measured by this questionnare
Children Functional Independence Measurement Scale | Before the intervention
  Functional Independency will be measured by this scale. Higher scores mean better independence.
Children Functional Independence Measurement Scale | After six weeks intervention
  Functional Independency will be measured by this scale. Higher scores mean better independence.
Lower extremity selective control measurement | Before the intervention
  Selective movement will be measured with this scale. Higher scores mean better selective control.
Lower extremity selective control measurement | After six weeks intervention
  Selective movement will be measured with this scale. Higher scores mean better selective control.

CONTACTS AND LOCATIONS:
Locations (1):
- Pelin Atalan, Izmir, Bornova, Turkey (Türkiye)